CLINICAL TRIAL: NCT05257278
Title: Single-center PMCF - Study on the Performance and Safety of MonoPlus® in Patients Undergoing Orthopedic Surgery
Brief Title: MonoPlus® in Orthopedic Surgery
Acronym: UNITE
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2027
Record Dates: First submitted 2022-02-17; First posted 2022-02-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Orthopedic Surgery; Soft Tissue Approximation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MonoPlus®: Patients undergoing orthopedic surgery with soft tissue approximation
  Interventions: Device: MonoPlus®

INTERVENTIONS:
Device: MonoPlus® — MonoPlus® is indicated for use in general soft tissue approximation, specially in cases where extended wound support of more than 4 weeks is desirable

SUMMARY:
Single-center postmarket clinical follow-up study (PMCF) on the performance and safety of MonoPlus® in patients undergoing orthopedic surgery

DETAILED DESCRIPTION:
This post-market clinical follow-up (PMCF) study on the use of MonoPlus®, a polydioxanone absorbable suture material, will expand the information available on the performance and safety of MonoPlus® used for orthopedic surgeries conducted in daily practice conditions.

The study is designed as a prospective, non-interventional, single-center, PMCF cohort study. The product under investigation will be used in routine clinical practice and according to the Instructions for Use. No diagnostic or therapeutic intervention outside of routine clinical practice will be applied, and all study visits will coincide with those that will be scheduled for routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Need for orthopedic surgery
* Use of MonoPlus® for the orthopedic surgery in the routine clinical practice
* Written informed consent form.

Exclusion Criteria:

* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to give informed consent and comply with the study procedures
* Prosthetic surgery secondary to infection
* Radiation to the surgical area
* Participation or planned participation in any clinical trial before study follow-up is completed
* Previous tendon/ligament repair intervention
* Pregnancy
* Patients with hypersensitivity or allergy to the suture material
* Patients taking medical consumption that might affect wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male of femal patients are eligible for inclusion in this study when they are in need of orthopedic surgery and MonoPlus® is used for soft tissue approximation for this orthopedic surgery in the routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Rate of maintained soft tissue approximation | 3 months post-surgery
  For the assessment of MonoPlus® effectiveness the percentage of patients that maintain soft tissue approximation integrity examined by ultrasound is evaluated

SECONDARY OUTCOMES:
Changes in functional performance for Patients undergoing Knee surgery | preoperatively, 6 weeks and 3 months post-surgery
  Mean changes in functional performance from baseline to week 6 and month 3 after surgery according to the Oxford Knee Score (OKS). OKS is a short 12-item patient-reported outcome(PRO) specifically designed and developed to assess function and pain with patients undergoing knee replacement surgery. When the OKS was originally developed, it was designed to be as simple as possible for ease of use. The scoring system is a 0-5 where one represented the best outcome. Item scores are summed to give a total score. The lower the score, the better the outcome.
Changes in functional performance for Patients undergoing Hip surgery | preoperatively, 6 weeks and 3 months post-surgery
  Mean changes in functional performance from baseline to week 6 and month 3 after surgery according to the Oxford Hip Score (OHS). The Oxford Hip Score (OHS) is a short 12-item patient-reported patient-reported outcome (PRO) specifically designed and developed to assess function and pain with patients undergoing hip replacement surgery. The OKS is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks. Each item has five possible responses from 0 to 5. Item scores are summed to give a total score. The lower the score, the better the outcome.
Changes in functional performance for Patients undergoing upper extremity surgery | preoperatively, 6 weeks and 3 months post-surgery
  Mean changes in functional performance from baseline to week 6 and month 3 after surgery according to the Quick Disability of Arm, Shoulder and Hand score (QuickDASH). The QuickDASH,is a subset of 11 items from the 30-item Disability of Arm, Shoulder and Hand score and is a self-reported questionnaire. The response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Changes in strength | at baseline, 6 weeks and 3 months post-surgery.
  Mean changes in strength measured by a dynamometer from baseline to week 6 and month 3 after surgery.
Incidence of reoperations | Up to last follow up 12 months post operatively
  Frequency of reoperation within the 12 months after surgery.
The length of hospital stay after the orthopedic surgery. | up to hospital discharge (approximately 10 days postoperatively)
  Mean duration of hospital stay in patients undergoing orthopedic surgery.
The incidence of post-surgery complicated wound healing. | 12-month study follow-up.
  Frequency of patients with complicated wound healing within the first 6 weeks post-surgery. A complicated wound healing will be recorded if the incision does not close completely, necrosis of the wound edge or primary or secondary dehiscence occur, or in cases of formation of a seroma, fistula, or bleeding.
The incidence of wound infections during the study follow-up. | 12-month study follow-up.
  Frequency of wound infections within the 12-month post-surgery follow-up. Wound infection is defined as redness, wound dehiscence with secretion (putrid or caliginous fluid), and / or microbiological evidence of bacterial contamination.
Development of Pain measured with Visual Analogue Scale (VAS) | Preoperatively, hospital discharge (approximately 10 days postoperatively), 6 weeks, 3 months and 12 months after surgery
  Mean pain VAS scores at rest and with activity at five different points of time (baseline, hospital discharge, 6 weeks, 3 months and 12 months after surgery. Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best).
Rate of Adverse Device Effects | up to last follow-up at 12 months postoperatively
  Frequencies of patients with Adverse Device Effects (ADE) reported until month 12 after surgery.
Assessment of intraoperative handling of suture material | intraoperatively
  Assessment of intraoperative handling of suture material using a questionnaire (Likert Scale) including various dimensions (knot security, tensile strength, knot run down, tissue drag and pliability) with 5 evaluation levels ('excellent' (5), 'very good' (4), 'good' (3), 'satisfied' (2) and 'poor' (1)).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sanz Ruiz, Principal Investigator — Gregorio Marañón Hospital
Locations (1):
- Hospital Gregorio Marañón, Madrid, Spain